CLINICAL TRIAL: NCT00950170
Title: AN OPEN-LABEL STUDY OF THE SAFETY AND EFFICACY OF REFACTO AF IN PREVIOUSLY UNTREATED PATIENTS IN USUAL CARE SETTINGS
Brief Title: Study of Safety And Efficacy Of ReFacto AF In Previously Untreated Hemophilia A Patients In The Usual Care Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3082B2-4434; B1831006 (Other: Alias Study Number); 2008-008436-93 (EudraCT Number)
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Hemophilia A
Keywords: ReFacto AF; factor VIII; inhibitors; antibodies
MeSH Terms: conditions — Hemophilia A | interventions — Clinical Laboratory Techniques; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The investigator treats subjects with ReFacto AF in the usual care setting.
  Interventions: Procedure: Laboratory Tests

INTERVENTIONS:
Procedure: Laboratory Tests — Blood draws to determine the level of factor VIII activity before and after dosing at appropriate visits, and blood draws to determine levels of factor VIII inhibitor (antibody to factor VIII).
  Other Names: ReFacto AF

SUMMARY:
Study to evaluate the safety and effectiveness of ReFacto AF for the treatment of severe hemophilia A in patients who have not yet received treatment for their hemophilia. Study subjects will be males less than 6 years old who have not taken any clotting factor or other blood products before the study. The safety and effectiveness of ReFacto AF will be determined in this study by tests and procedures done at the doctor's office.

DETAILED DESCRIPTION:
Regulatory Commitment

ELIGIBILITY:
Inclusion Criteria:

* Male subjects <6 years of age with severe hemophilia A (FVIII:C <1%) based on clinical records, including newborns.
* No prior exposure to factor products or any blood products.

Exclusion Criteria:

* Presence of any bleeding disorder in addition to hemophilia A.
* Treatment with any investigational agent or device within the past 30 days.
* Any condition(s) that compromises the ability to collect study-related observations, or that poses a contraindication to study participation (these conditions include, but are not limited to, inadequate medical history to assure study eligibility; and expectation of poor adherence to study requirements).

Max Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2010-02-10 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- CHU de Nantes, Nantes, France
- Germany (2):
  - Medizinische Hochschule, Hannover, Hanover, Lower Saxony
  - Klinikum Bremen-Mitte gGmbH, Professor Hess Kinderklinik, Bremen
- Agenzia per L'emofilia e Centro Regionale Riferimento Coagulopatie Congenite, Florence, Italy
- University Medical Center Groningen, Groningen, Netherlands
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Fe, Valencia
- Turkey (Türkiye) (3):
  - Ege Universitesi Tip Fakultesi, Bornova, İzmir
  - Cukurova Universitesi Tip Fakultesi, Adana
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
- Derzhavna ustanova "Instytut patolohii krovi ta transfuziinoi medytsyny Natsionalnoi akademii, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-4434&StudyName=Study%20of%20Safety%20And%20Efficacy%20Of%20ReFacto%20AF%20In%20Previously%20Untreated%20Hemophilia%20A%20Patients%20In%20The%20Usual%20Care%20Setting

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 participants were enrolled in this non-randomized open-label study & they received ReFacto albumin free (AF) at dose & frequency prescribed by each participant's treating physician as per local standard of care & in accordance with summary of product characteristics (SmPC). Participants were expected to be in study for about 26 months
Pre-assignment Details: The study was conducted at 11 centers across various countries. Participants less than 6 years of age with severe hemophilia A (FVIII activity in plasma [FVIII:C]<1%) who had not received any prior factor products or blood products for their hemophilia A were enrolled in this study.
Groups:
- Overall Participants: All participants enrolled in the study who had received at least 1 dose of ReFacto AF.
Period: Overall Study
Arm/Group | Overall Participants
Started | 23
Completed | 19
Not Completed | 4
Not completed — Parent/Legal Guardian Request | 1
Not completed — Adverse Event | 2
Not completed — Discontinuation of Study by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who took at least 1 dose of study medication.
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.0 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Clinically Significant Factor VIII (FVIII) Inhibitors During the Course of the Study
Description: Percentage of participants who developed clinically significant FVIII inhibitors: those persistent over a defined period with clinically impactful effects like breakthrough bleed, low recovery, etc., during the course of the study.
Time Frame: 2 years
Population: Analysis set included all participants who had received at least 1 dose of ReFacto AF and those were observed for clinically significant FVIII inhibitors.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
Percentage of participants | 21.74 [7.46 to 43.70]

2. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: Annualized bleeding rate was calculated as the number of bleeds divided by the treatment interval duration (enrollment visit to final visit) and then multiplied by 365.25. If there was more than 1 bleed location (like ankle and joint) with identical bleed start date and time, it was treated as 1 bleed occurrence.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
bleeds per year | 5.88 (8.082)

3. Secondary Outcome: Total Number of Infusions to Treat a New Bleed Classified on Basis of Response to First On-Demand Treatment With Refacto AF
Description: Number of infusions of Refacto AF required to treat a new bleed were classified on basis of the response to at 4-point response scale of assessment (excellent, good, moderate and no response). Assessment was completed each time a participant experienced a new bleed requiring an 'on-demand' IV infusion. Excellent: definite pain relief and/or improvement in bleeding signs within 8 hours (hr) after infusion, no additional infusion administered; Good: definite pain relief and/or improvement in bleeding signs within 8 hr after infusion, at least 1 additional infusion administered for complete resolution or with no additional infusion administered; Moderate: probable or slight improvement starting after 8 hr following infusion, at least 1 additional infusion administered for complete resolution; No Response: no improvement at all between infusions or during 24 hr interval following infusion or condition worsen. Bleeds for which response not recorded, reported as: Data Not Recorded.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Groups:
- Overall Participants: First IV Infusion Per Bleed: First IV infusions of ReFacto AF received by the participants for on-demand treatment of new bleed.
- Overall Participants: Follow-up IV Infusions: Follow-up IV infusions of ReFacto AF received by the participants for on-demand treatment of new bleed.
- Overall Participants: All IV Infusions: A sum of all IV infusions of ReFacto AF received by the participants for on-demand treatment of new bleed.
Arm/Group | Overall Participants: First IV Infusion Per Bleed | Overall Participants: Follow-up IV Infusions | Overall Participants: All IV Infusions
Number analyzed (Participants) | 23 | 23 | 23
Number analyzed (Infusions) | 149 | 44 | 193
Infusions
  Excellent | 51 | 7 | 58
  Good | 48 | 19 | 67
  Moderate | 28 | 12 | 40
  No response | 3 | 5 | 8
  Data not recorded | 19 | 1 | 20

4. Secondary Outcome: Total Number of Infusions Needed for Resolution of Bleeding Episodes Classified on Basis of Response to Study Drug Infusion
Description: Number of infusions of Refacto AF required for resolution of a bleeding episodes were classified on basis of the response at 4-point response scale of assessment (excellent, good, moderate and no response). Excellent: definite pain relief and/or improvement in bleeding signs within 8 hours (hr) after infusion, no additional infusion administered; Good: definite pain relief and/or improvement in bleeding signs within 8 hr after infusion, at least 1 additional infusion administered for complete resolution or with no additional infusion administered; Moderate: probable or slight improvement starting after 8 hr following infusion, at least 1 additional infusion administered for complete resolution; No Response: no improvement at all between infusions or during 24 hr interval following infusion or condition worsen. Bleeds for which response not recorded, reported as: Data Not Recorded.
Time Frame: Within 48 hours after infusion, up to 2 years treatment duration
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Groups:
- One IV Infusion: One IV infusion of ReFacto AF received by the participants.
- Two IV Infusions: Two IV infusions of ReFacto AF received by the participants.
- Three IV Infusions: Three IV infusions of ReFacto AF received by the participants.
- Four IV Infusions: Four IV infusions of ReFacto AF received by the participants.
- Greater Than 4 IV Infusions: > 4 IV infusions of ReFacto AF received by the participants.
- Total Number of Bleeds: Total number of bleeds reported in the study.
Arm/Group | One IV Infusion | Two IV Infusions | Three IV Infusions | Four IV Infusions | Greater Than 4 IV Infusions | Total Number of Bleeds
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
Number analyzed (Infusions) | 132 | 13 | 1 | 0 | 4 | 150
Infusions
  Excellent | 48 | 3 | 0 |  | 0 | 51
  Good | 43 | 5 | 0 |  | 1 | 49
  Moderate | 22 | 4 | 0 |  | 2 | 28
  No response | 2 | 0 | 0 |  | 1 | 3
  Data Not Recorded | 17 | 1 | 1 |  | 0 | 19

5. Secondary Outcome: Total Number of Breakthrough Bleeding Episodes Occurring Within 48 Hours After a Prophylaxis Infusion of ReFacto AF
Description: The number of breakthrough bleeds (spontaneous or traumatic) within 48 hours following a prophylaxis dose of ReFacto AF are summarized. If there was more than 1 bleed location (like ankle and joint) with identical bleed start date and time, it was treated as 1 bleed occurrence.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Number; unit: Bleeding episodes
Groups:
- Overall Participants: Breakthrough Bleeds: All participants enrolled in the study who received at least 1 dose of ReFacto AF and had a bleeding episode within 48 hours after a prophylaxis infusion of ReFacto AF.
Arm/Group | Overall Participants: Breakthrough Bleeds
Number analyzed (Participants) | 9
Bleeding episodes | 12

6. Secondary Outcome: Consumption of Total International Units of Factor VIII
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: International units
Groups:
- Overall Participants: On Demand: All participants enrolled in the study who received at least 1 dose of ReFacto AF in on demand setting.
- Overall Participants: Preventive: All participants enrolled in the study who received at least 1 dose of ReFacto AF in preventive setting.
- Overall Participants: Prophylaxis: All participants enrolled in the study who received at least 1 dose of ReFacto AF in prophylaxis setting.
- Overall Participants: Setting Not Specified: All participants enrolled in the study who received at least 1 dose of ReFacto AF in unspecified setting.
- Overall Participants: All participants enrolled in the study who received at least 1 dose of ReFacto AF.
Arm/Group | Overall Participants: On Demand | Overall Participants: Preventive | Overall Participants: Prophylaxis | Overall Participants: Setting Not Specified | Overall Participants
Number analyzed (Participants) | 21 | 7 | 22 | 4 | 23
International units | 4186 (3038.4) | 1857 (2357.5) | 55543 (55535.5) | 1634 (2523.8) | 57799 (55125.8)

7. Secondary Outcome: Consumption of Total International Units of Factor VIII Per Year
Description: Consumption of total international units of Factor VIII per year was calculated for a participant: dividing the total consumption of factor VIII by participant's treatment interval duration (in days), then multiplying by 365.25.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
International units per year | 72336 (123407.9)

8. Secondary Outcome: Mean Dose (IU) of Study Drug Consumed Per Infusion
Description: Mean dose for each participant was calculated as participant's total factor VIII consumption (in IU) divided by the number of infusions administered.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: International units per infusion
Arm/Group | Overall Participants: On Demand | Overall Participants: Preventive | Overall Participants: Prophylaxis | Overall Participants: Setting Not Specified | Overall Participants
Number analyzed (Participants) | 21 | 7 | 22 | 4 | 23
International units per infusion | 552 (296.7) | 544 (285.6) | 628 (389.6) | 481 (401.5) | 619 (386.5)

9. Secondary Outcome: Consumption of Total International Units of Factor VIII by Weight
Description: Consumption of total international units of Factor VIII by weight was calculated for a participant: dividing the total consumption of factor VIII by participant's weight (the most recently recorded).
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: International units per kilogram
Arm/Group | Overall Participants: On Demand | Overall Participants: Preventive | Overall Participants: Prophylaxis | Overall Participants: Setting Not Specified | Overall Participants
Number analyzed (Participants) | 21 | 7 | 22 | 4 | 23
International units per kilogram | 388 (297.0) | 93 (56.8) | 4766 (4933.5) | 187 (256.5) | 4966 (4891.4)

10. Secondary Outcome: Consumption of Total International Units of Factor VIII Per Year by Weight
Description: Consumption of total international units of Factor VIII per year by weight was calculated for a participant: the total consumption of factor VIII divided by participant's treatment interval duration (in days), then multiplying by 365.25 and then dividing by participant's weight (the most recently recorded).
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: International units per kilogram*years
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
International units per kilogram*years | 6398 (11102.8)

11. Secondary Outcome: Mean Dose (IU) of Study Drug Consumed Per Infusion by Weight
Description: Mean dose for each participant was calculated as participant's total factor consumption (in IU) divided by the number of infusions administered and then dividing by participant's weight (the most recently recorded).
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: International units per kilogram
Arm/Group | Overall Participants: On Demand | Overall Participants: Preventive | Overall Participants: Prophylaxis | Overall Participants: Setting Not Specified | Overall Participants
Number analyzed (Participants) | 21 | 7 | 22 | 4 | 23
International units per kilogram | 49 (26.1) | 42 (16.9) | 55 (34.4) | 50 (41.0) | 53 (33.5)

12. Secondary Outcome: Mean of Total Number of Infusions of Study Drug Received
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Overall Participants: On Demand | Overall Participants: Preventive | Overall Participants: Prophylaxis | Overall Participants: Setting Not Specified | Overall Participants
Number analyzed (Participants) | 21 | 7 | 22 | 4 | 23
Infusions | 9 (8.0) | 5 (8.9) | 80 (36.9) | 2 (1.9) | 86 (37.5)

13. Secondary Outcome: Mean of Total Number of Days Participants Exposed to Study Drug
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Overall Participants: On Demand | Overall Participants: Preventive | Overall Participants: Prophylaxis | Overall Participants: Setting Not Specified | Overall Participants
Number analyzed (Participants) | 21 | 7 | 22 | 4 | 23
Days | 8 (6.3) | 3 (3.7) | 76 (31.3) | 2 (1.9) | 81 (32.4)

14. Secondary Outcome: Number of Participants Who Required Dose Escalation of Their Prescribed Prophylaxis Regimen During Their Participation in This Study
Description: The number of participants who met the dose escalation criteria were prescribed a higher dose and/or were prescribed more frequent doses. When dose escalation was required, the specific dose and dosing schedule was at the investigator's discretion.
Time Frame: 2 years
Population: Efficacy analysis set consisted of all participants who had received at least 1 dose of ReFacto AF.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Participants: Prophylaxis
Number analyzed (Participants) | 22
Participants | 15

15. Secondary Outcome: Percentage of Bleeding Episodes With Less-Than-Expected Therapeutic Effect (LETE) in On-Demand (OD) Setting
Description: LETE occurs in OD setting if participant recorded 2 successive "No Response" (no improvement at all between infusions, or condition worsens) ratings after 2 successive infusions of study drug. Infusions must have been given within 24 hours (hr) of each other for treatment of same bleeding event in absence of confounding factors (known presence or subsequent identification of a FVIII inhibitor, known inadequate dose for type and/or severity of bleed in opinion of investigator, delay of greater than (>) 4 hr between onset of bleed to infusion, delay of >24 hr before administration of a follow-up infusion, known compromised study drug, faulty administration of study drug, participant had an underlying, predisposing condition responsible for bleed in opinion of investigator, ongoing trauma responsible for continued bleeding.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Number (95% Confidence Interval); unit: Percentage of bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
Number analyzed (Bleeding episodes) | 150
Percentage of bleeding episodes | 0 [0.00 to 2.43]

16. Secondary Outcome: Percentage of Bleeding Episodes With Less-Than-Expected Therapeutic Effect (LETE) in the Prophylaxis Setting
Description: LETE in prophylaxis setting if there was a spontaneous bleed within 48 hours after a regularly scheduled prophylactic dose of study drug (which was not used to treat a bleed) in the absence of confounding factors (known presence or subsequent identification of a FVIII inhibitor, known inadequate prophylactic dose [a dose less than that prescribed in participant's regimen], known lack of adherence to the prescribed prophylaxis regimen, known compromised study drug, faulty administration of study drug, participant had an underlying, predisposing condition responsible for the bleed in the opinion of the investigator, traumatic injury responsible for bleeding.
Time Frame: 2 years
Population: Efficacy analysis set included all participants who had received at least 1 dose of ReFacto AF.
Measure: Number (95% Confidence Interval); unit: Percentage of bleeding episodes
Units Other Than Participants: Routine prophylaxis infusions
Arm/Group | Overall Participants: Prophylaxis
Number analyzed (Participants) | 22
Number analyzed (Routine prophylaxis infusions) | 1752
Percentage of bleeding episodes | 0.11 [0.01 to 0.41]

17. Secondary Outcome: Total Number of Events of Potential Less-Than-Expected Therapeutic Effect (LETE) in the Low Recovery Setting
Description: LETE was lower than expected recovery of FVIII in the opinion of the investigator following infusion of study drug in the absence of confounding factors (known presence or subsequent identification of a FVIII inhibitor, known compromised study drug, faulty administration of study drug including inadequate dosing).
Time Frame: 2 years
Population: Efficacy analysis set consisted of all participants who had received at least 1 dose of ReFacto AF.
Measure: Number; unit: Events
Groups:
- Overall Participants: All participants who received at least 1 dose of ReFacto AF.
Arm/Group | Overall Participants
Number analyzed (Participants) | 23
Events | 10

ADVERSE EVENTS:
Time Frame: Through study completion up to 2 years
Description: Event may be serious in 1 and non serious in other participant or 1 participant may have experienced both serious and non serious adverse event.
Arm/Group | Overall Participants
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Participants (N=23)
Appendicitis (Infections and infestations) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1)
Milk allergy (Immune system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Factor VIII inhibition (Blood and lymphatic system disorders) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Participants (N=23)
Gastroenteritis (Infections and infestations) | 6 (7)
Nasopharyngitis (Infections and infestations) | 6 (14)
Bronchitis (Infections and infestations) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Conjunctivitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (3)
Rhinitis (Infections and infestations) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Teething (Gastrointestinal disorders) | 2 (3)
Pyrexia (General disorders) | 10 (13)
Fall (Injury, poisoning and procedural complications) | 4 (8)
Head injury (Injury, poisoning and procedural complications) | 2 (3)
Lip injury (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 (5)
Haematoma (Vascular disorders) | 4 (5)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator may publish or otherwise publicly communicate the results, subject to the provisions of the Clinical Study Agreement.